CLINICAL TRIAL: NCT05670444
Title: Melatonin, Vitamins and Minerals Supplements for the Treatment of Covid-19 and Covid-like Illness: Results of a Prospective, Randomised, Double-blinded Multicentre Study
Brief Title: Melatonin, Vitamins and Minerals Supplements for the Treatment of Covid-19 and Covid-like Illness
Acronym: kela-cov
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hôpital Universitaire Sahloul (Other)
Responsible Party: Principal Investigator, Riadh Boukef, chef of emergency departement, Hôpital Universitaire Sahloul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: kelavit
Record Dates: First submitted 2022-12-26; First posted 2023-01-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Influenza -Like Illness

STUDY DESIGN:
Intervention Model Description: multicenter, randomized , placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kelavit (Active Comparator): The treatment group received two pills in the morning containing Vit C Vit D zinc and minerals and one pill of 2 mg of melatonin in the evening
  Interventions: Drug: kelavit
- placebo (Placebo Comparator): Patients from the placebo group received three similar pills
  Interventions: Drug: kelavit

INTERVENTIONS:
Drug: kelavit — The treatment group received two pills in the morning containing Vit C Vit D zinc and minerals and one pill of 2 mg of melatonin in the evening

SUMMARY:
a multicenter, double-blind, randomized, placebo-controlled trial. Patients aged less than 60 years old with no previous medical history consulting the emergency department for covid and covid-like illness and who were not hospitalized were included. Those who have known allergy or severe side effect on the study drugs and those who refused to consent were excluded. Pregnant women were not included. For all the included patients, a PCR test for the detection of SARS COV2 was realized. Patients were assigned in a 1:1 ratio to the treatment group or the placebo group. The treatment group received two pills in the morning containing Vit C Vit D zinc and minerals and one pill of 2 mg of melatonin in the evening . Patients from the placebo group received three similar pills . The pills were identical in color, taste, smell, consistency, and container

DETAILED DESCRIPTION:
This was a multicenter, double-blind, randomized, placebo-controlled trial. The study was approved by the ethics committee of the the Faculty of Medicine "Ibn El Jazzar" of Sousse. Patients provided written informed consent before participation. Patients were recruited from Sahloul emergency department, F.Hached emergency department, F.Bourguiba emergency department. Patients aged less than 60 years old with no previous medical history consulting the emergency department for covid and covid-like illness and who were not hospitalized were included. Those who have known allergy or severe side effect on the study drugs and those who refused to consent were excluded. Pregnant women were not included. For all the included patients, a PCR test for the detection of SARS COV2 was realized. Patients were assigned in a 1:1 ratio to the treatment group or the placebo group. The randomization list was created using a computer-generated code. A staff member who had no role in the study managed the randomization. The treatment group received two pills in the morning containing Vit C Vit D zinc and minerals and one pill of 2 mg of melatonin in the evening . Patients from the placebo group received three similar pills . The pills were identical in color, taste, smell, consistency, and container. They were prepared by XEn Plus laboratory members and labeled by a staff member who did not participate in the study. Patients and investigators remained blinded to randomization until the final analysis. After consenting, patients were examined by an emergency resident. They were asked about the common Covid-19 and Covid-like illness signs: fever, headache, asthenia/fatigue, sputum expectoration, anosmia, chills, skin rash, diarrhea, sore throat, abdominal pain, cough, vomiting, chest pain, hemoptysis, joint pain, ageusia, dyspnea, muscle pain and conjunctives. On physical examination vital signs were checked: blood pressure, pulse rate, respiration rate, body temperature, glycemic index, oxygen saturation and height and weight. This symptoms were assessed using a scale from 0 to 3 (not at all, slight, a lot, awful) and they were monitored via telecommunication. A follow-up was carried for each included patient on day 1, day 10, day 15 and day 30. Compliance with treatment, the date of disappearance of symptoms, side effects, adverse events, hospitalization, respiratory assistance requirement and death were mentioned accordingly

ELIGIBILITY:
Inclusion Criteria:

* Patients aged less than 60 years old
* no previous medical history
* consulting the emergency department for covid and covid-like illness
* not hospitalized

Exclusion Criteria:

* allergy or severe side effect on the study drugs
* refused to consent
* Pregnant women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
mortality rate | 30 days after inclusion
  death rate
need for ICU admission | 30 days after inclusion
  Number of participants admitted to the intensive care unit
combined outcome | 30 days after inclusion
  death or need for admission to the ICU for COVID-19 related complications

SECONDARY OUTCOMES:
Date of disappearance of symptoms present on admission | 30 days after inclusion
  Date of disappearance of symptoms present on admission
appearance of an adverse effect due to the administration of the treatment | 30 days after inclusion
  appearance of an adverse effect due to the administration of the treatment
number of patients developing complications | 30 days after inclusion
  number of patients developing complications
number of participants requiring hospitalization due to COVID- infection | 30 days after inclusion
  number of participants requiring hospitalization due to COVID- infection
number of participants requiring respiratory support or hospitalization | 30 days after inclusion
  number of participants requiring respiratory support or hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU sahloul, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No
in the article publication